CLINICAL TRIAL: NCT03493113
Title: Transient Hypothyroxinemia of Prematurity: Electrophysiological Changes in the Preterm Infants' Brain, a Retrospective Study
Brief Title: EEG Alterations in Preterm Infants With Thyroid Dysfunction
Acronym: EEG-THOP
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S61028
Record Dates: First submitted 2017-11-27; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2017-11

CONDITIONS: Transient Hypothyroxinemia of Prematurity
Keywords: EEG
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: EEG

SUMMARY:
The aim of this study is to investigate differences in electroencephalography (EEG) evolution between preterm infants with and without transient hypothyroxinemia of prematurity (THOP) in order to find differences in the interburst interval and the background pattern and in the maturation of the sleep-wake cycle.

DETAILED DESCRIPTION:
1. Definition of THOP The determination of thyroid hormones (TH) are assay-specific and related to the infants' gestational age (GA) and moment of determination. Immediately after birth, there will be a surge of TH, subsequently followed by a decrease to basal levels. Therefore, it is difficult to obtain reference values.

   The investigators plan to set out specific reference values for the preterm patient population, based on the TH laboratory results of cord blood, performed in the clinical laboratory of UZ Leuven and available over the last 4 years. The results will be linked to the gestational age. Dependent whether the data distribution is normal or not, the investigators are planning to use standard deviations or percentiles to classify patients.
2. EEG findings In this retrospective study, quantitative EEG- sleep behavior at (near) term age (GA 36-44 weeks) in preterm infants born <28 weeks GA, will be analyzed (n = 87).

EEGs were taken in the framework of the Resilience study and hereby, parental informed consent was already obtained.

TH function is assessed in preterm infants ≤ 34 weeks as part of the clinical care protocol. No additional blood samples were taken.

Quantitative EEG measures will be compared between the preterm infants with THOP (circulating thyroxine levels< P10) and without THOP. Logisitic regression will be performed to determine the effect of thyroid function as well as other clinical and demographic variables, on functional brain development at term equivalent age. These results will also be linked to long-term neurodevelopment outcome.

In a subgroup of these preterm patients (n=42) sequential EEGs, recorded during their stay at the neonatal intensive care unit, are available. These EEGs will be analyzed in a fully automatic way to assess functional EEG- brain maturation.

In this way, the investigators want to investigate whether deviations of normal preterm EEG-brain maturation can be discerned in preterm neonates with THOP and without THOP.

In preterm infants with GA < 32 weeks, developmental follow up data are available at the corrected age of 9 months and 2 years (Follow up Convention). The investigators will use these results and link them to the EEG findings and THOP data.

ELIGIBILITY:
Inclusion Criteria:

* gestational age < 28 weeks
* serial EEG recordings available
* thyroid function test on the first day of life and at the end of the first week of life available

Exclusion Criteria:

* Presence of congenital abnormalities

Ages: 24 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants who had EEG recordings in the framework of the Resilience study and gestational age < 28 weeks.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Differences in EEG measures in preterm infants with thyroid dysfunction | November 2011 - November 2017
  Quantitative EEG measures will be compared between the preterm infants with THOP (circulating T4 level< P10) and without THOP. In a subgroup of these preterm patients (n=42) sequential EEGs, recorded during their stay at the NICU, are available. These EEGs will be analyzed in a fully automatic way to assess functional EEG- brain maturation.

SECONDARY OUTCOMES:
Neurodevelopmental disturbances due to THOP and predicted by EEG alterations | November 2011 - November 2019
  In preterm infants with GA < 32 weeks, developmental follow up data are available at the corrected age of 9 months and 2 years (Follow up Convention). We will use these results and link them to the EEG findings and THOP data.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Department of Neonatology, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] La Gamma EF, Paneth N. Clinical importance of hypothyroxinemia in the preterm infant and a discussion of treatment concerns. Curr Opin Pediatr. 2012 Apr;24(2):172-80. doi: 10.1097/MOP.0b013e32835067cc. PMID 22273635
- [Result] Reuss ML, Paneth N, Pinto-Martin JA, Lorenz JM, Susser M. The relation of transient hypothyroxinemia in preterm infants to neurologic development at two years of age. N Engl J Med. 1996 Mar 28;334(13):821-7. doi: 10.1056/NEJM199603283341303. PMID 8596548
- [Result] Leviton A, Paneth N, Reuss ML, Susser M, Allred EN, Dammann O, Kuban K, Van Marter LJ, Pagano M. Hypothyroxinemia of prematurity and the risk of cerebral white matter damage. J Pediatr. 1999 Jun;134(6):706-11. doi: 10.1016/s0022-3476(99)70285-4. PMID 10356138
- [Result] Auso E, Lavado-Autric R, Cuevas E, Del Rey FE, Morreale De Escobar G, Berbel P. A moderate and transient deficiency of maternal thyroid function at the beginning of fetal neocorticogenesis alters neuronal migration. Endocrinology. 2004 Sep;145(9):4037-47. doi: 10.1210/en.2004-0274. Epub 2004 Apr 15. PMID 15087434
- [Result] Santisteban P, Bernal J. Thyroid development and effect on the nervous system. Rev Endocr Metab Disord. 2005 Aug;6(3):217-28. doi: 10.1007/s11154-005-3053-9. No abstract available. PMID 16151626
- [Result] Fisher DA. Thyroid system immaturities in very low birth weight premature infants. Semin Perinatol. 2008 Dec;32(6):387-97. doi: 10.1053/j.semperi.2008.09.003. PMID 19007675
- [Result] Shellhaas RA, Burns JW, Barks JD, Chervin RD. Quantitative sleep stage analyses as a window to neonatal neurologic function. Neurology. 2014 Feb 4;82(5):390-5. doi: 10.1212/WNL.0000000000000085. Epub 2014 Jan 2. PMID 24384644
- [Result] Scher MS, Loparo KA. Neonatal EEG/sleep state analyses: a complex phenotype of developmental neural plasticity. Dev Neurosci. 2009;31(4):259-75. doi: 10.1159/000216537. Epub 2009 Jan 2. PMID 19546563
- [Result] Koolen N, Dereymaeker A, Rasanen O, Jansen K, Vervisch J, Matic V, Naulaers G, De Vos M, Van Huffel S, Vanhatalo S. Early development of synchrony in cortical activations in the human. Neuroscience. 2016 May 13;322:298-307. doi: 10.1016/j.neuroscience.2016.02.017. Epub 2016 Feb 11. PMID 26876605
- [Result] Shellhaas RA, Burns JW, Hassan F, Carlson MD, Barks JDE, Chervin RD. Neonatal Sleep-Wake Analyses Predict 18-month Neurodevelopmental Outcomes. Sleep. 2017 Nov 1;40(11):zsx144. doi: 10.1093/sleep/zsx144. PMID 28958087
- [Result] Scher MS, Steppe DA, Banks DL. Prediction of lower developmental performances of healthy neonates by neonatal EEG-sleep measures. Pediatr Neurol. 1996 Feb;14(2):137-44. doi: 10.1016/0887-8994(96)00013-6. PMID 8703226
- [Result] Niemarkt HJ, Jennekens W, Maartens IA, Wassenberg T, van Aken M, Katgert T, Kramer BW, Gavilanes AW, Zimmermann LJ, Bambang Oetomo S, Andriessen P. Multi-channel amplitude-integrated EEG characteristics in preterm infants with a normal neurodevelopment at two years of corrected age. Early Hum Dev. 2012 Apr;88(4):209-16. doi: 10.1016/j.earlhumdev.2011.08.008. Epub 2011 Sep 15. PMID 21924567
- [Result] Niemarkt HJ, Jennekens W, Pasman JW, Katgert T, Van Pul C, Gavilanes AW, Kramer BW, Zimmermann LJ, Bambang Oetomo S, Andriessen P. Maturational changes in automated EEG spectral power analysis in preterm infants. Pediatr Res. 2011 Nov;70(5):529-34. doi: 10.1203/PDR.0b013e31822d748b. PMID 21772227
- [Result] Khedr EM, El Toony LF, Tarkhan MN, Abdella G. Peripheral and central nervous system alterations in hypothyroidism: electrophysiological findings. Neuropsychobiology. 2000 Jan;41(2):88-94. doi: 10.1159/000026638. PMID 10644929
- [Result] Fisher DA, Odell WD. Acute release of thyrotropin in the newborn. J Clin Invest. 1969 Sep;48(9):1670-7. doi: 10.1172/JCI106132. PMID 5822577
- [Result] Williams FL, Simpson J, Delahunty C, Ogston SA, Bongers-Schokking JJ, Murphy N, van Toor H, Wu SY, Visser TJ, Hume R; Collaboration from the Scottish Preterm Thyroid Group. Developmental trends in cord and postpartum serum thyroid hormones in preterm infants. J Clin Endocrinol Metab. 2004 Nov;89(11):5314-20. doi: 10.1210/jc.2004-0869. PMID 15531476
- [Result] Dereymaeker A, Pillay K, Vervisch J, Van Huffel S, Naulaers G, Jansen K, De Vos M. An Automated Quiet Sleep Detection Approach in Preterm Infants as a Gateway to Assess Brain Maturation. Int J Neural Syst. 2017 Sep;27(6):1750023. doi: 10.1142/S012906571750023X. Epub 2017 Feb 24. PMID 28460602
- [Result] Stevenson NJ, Oberdorfer L, Koolen N, O'Toole JM, Werther T, Klebermass-Schrehof K, Vanhatalo S. Functional maturation in preterm infants measured by serial recording of cortical activity. Sci Rep. 2017 Oct 11;7(1):12969. doi: 10.1038/s41598-017-13537-3. PMID 29021546
- [Result] Dereymaeker A, Koolen N, Jansen K, Vervisch J, Ortibus E, De Vos M, Van Huffel S, Naulaers G. The suppression curve as a quantitative approach for measuring brain maturation in preterm infants. Clin Neurophysiol. 2016 Aug;127(8):2760-2765. doi: 10.1016/j.clinph.2016.05.362. Epub 2016 Jun 8. PMID 27417049